CLINICAL TRIAL: NCT03184571
Title: A Phase II Multi Center Study of BGB324 in Combination With Pembrolizumab in Patients With Previously Treated Advanced Adenocarcinoma of the Lung
Brief Title: Bemcentinib (BGB324) in Combination With Pembrolizumab in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGBC008; MK-3475 PN531 (Other: MSD); 2016-003609-32 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer Metastatic; NSCLC Stage IV; Adenocarcinoma of Lung
Keywords: bemcentinib; NSCLC; pembrolizumab; Keytruda; BGB324
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — pembrolizumab; bemcentinib

STUDY DESIGN:
Intervention Model Description: Extension to Simon's 2-stage design allowing termination at the end of Stage 1 for either futility or efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A Bemcentinib + pembrolizumab (Experimental): Cohort A bemcentinib (BGB324) in combination with pembrolizumab will be administered to participants with previously treated, advanced adenocarcinoma of the lung who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy.
  Interventions: Drug: Pembrolizumab; Drug: Bemcentinib
- Cohort B Bemcentinib + pembrolizumab (Experimental): Cohort B bemcentinib (BGB324) in combination with pembrolizumab will be administered to participants with previously treated, advanced adenocarcinoma of the lung who received a maximum of one prior line of an anti-PD-(L)1 therapy (monotherapy).
  Interventions: Drug: Pembrolizumab; Drug: Bemcentinib
- Cohort C Bemcentinib + pembrolizumab (Experimental): Cohort C bemcentinib (BGB324) in combination with pembrolizumab will be administered to participants with previously treated, advanced adenocarcinoma of the lung who received a maximum of one prior line of therapy with an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy.
  Interventions: Drug: Pembrolizumab; Drug: Bemcentinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a PD-1 inhibitor
  Other Names: Keytruda
Drug: Bemcentinib — Bemcentinib is a selective Axl kinase inhibitor;
  Other Names: BGB324

SUMMARY:
This is an open-label, multi-center, single arm, phase II study to assess the anti-tumor activity and safety of bemcentinib in combination with pembrolizumab in up to 106 participants with previously treated, advanced adenocarcinoma of the lung. The study will enrol three cohorts of participants with previously treated, advanced adenocarcinoma of the lung. Cohort A will consist of participants who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy. Cohort B will consist of participants who received a maximum of one prior line of an anti-programmed death receptor (PD)-(L)1 therapy (monotherapy). Cohort C will consist of participants who received a maximum of one prior line of therapy with an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy. The primary objective is to assess the anti-tumor activity of bemcentinib in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent.
2. Male and non-pregnant females who were aged 18 years or older at the time of provision of informed consent.
3. Histopathologically or cytologically documented Stage IV adenocarcinoma NSCLC; Note: Patients with a mixed cell histology including a significant area of adenocarcinoma histology were eligible.
4. Cohort A: Had disease progression on or after a prior platinum-containing chemotherapy; Note: Patients with EGFR mutations or ALK genomic rearrangements had to have documented disease progression on at least 1 licensed therapy for these indications and may not have received platinum-containing chemotherapy.

   Cohort B:
   1. Had received a maximum of 1 prior line of an anti-PD-(L)1 therapy (monotherapy).
   2. Must have had disease control containing at least 2 doses of anti-PD-(L)1 therapy. Disease control was defined as:

   i. Stable disease for at least 12 weeks (date of first progression on anti-PD-(L)1 therapy) Or ii. Confirmed PR or CR - confirmatory scan must have been performed >4 weeks from initial scan) c) Had disease progression when entering Screening (first date of progression of disease was taken as end date of response to previous anti-PD-(L)1 therapy) and this must have been within 12 weeks of last dose of treatment containing an anti-PD-(L)1 therapy. Progression should have been confirmed in 1 of the following ways: i. Having had 2 scan assessments completed at least 4 weeks apart, both showing progression according to response evaluation criteria in solid tumors (RECIST) 1.113 or ii. Having had 1 scan assessment completed showing disease progression according to standards used for previous therapy combined with rapid disease progression / clinical progression.

   Cohort C:
   1. Had received a maximum of 1 prior line of an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy.
   2. Must have had disease control containing at least 2 doses of anti-PD-(L)1 therapy. Disease control was defined as:

   i. Stable disease for at least 12 weeks (date of first progression on anti-PD-(L)1 therapy) Or ii. Confirmed PR or CR - confirmatory scan must be performed >4 weeks from initial scan c) Had disease progression when entering Screening (first date of progression of disease was taken as end date of response to previous anti-PD-(L)1 therapy) and this must have been within 12 weeks of last dose of treatment containing an anti-PD-(L)1 therapy. Progression had to be confirmed in 1 of the following ways: i. Having had 2 scan assessments completed at least 4 weeks apart, both showing progression according to RECIST 1.113 or ii. Having had 1 scan assessment completed showing disease progression according to standards used for previous therapy combined with rapid disease progression/clinical progression
5. Measurable disease as defined by RECIST 1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) and as determined by the site study team; tumor lesions situated in a previously irradiated area were considered measurable if progression had been demonstrated in such lesions.
6. Provision of suitable tumor tissue for the analysis of AXL kinase expression and PD-L1 expression; suitable tumor tissue had to consist of a minimum of a newly acquired (fresh) tumor tissue sample (as a formalin-fixed paraffin-embedded [FFPE] block), together with either further newly acquired tumor tissue (ie, further FFPE block) or an archival tumor tissue sample (as a further FFPE block or further 10 unstained slides).
7. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
8. Life expectancy of at least 3 months
9. Adequate organ function confirmed at Screening within 10 days of treatment initiation as evidenced by:

   1. Platelet count ≥100,000/mm3
   2. Hemoglobin ≥9.0 g/dL (≥5.6 mmol/L)
   3. Absolute neutrophil count >1,500/mm3
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × the upper limit of normal (ULN), or ≤5 × the ULN for patients with liver metastases
   5. Total bilirubin ≤1.5 × the ULN, or direct bilirubin < ULN for patients with total bilirubin levels >1.5 ULN
   6. Creatinine ≤1.5 × the ULN or calculated creatinine clearance 60 mL/min (by Cockcroft Gault formula)
   7. International normalized ratio or prothrombin time ≤1.5 × the ULN and activated partial thromboplastin time ≤1.5 × the ULN; Note: If patient was receiving anticoagulant therapy, then prothrombin time or partial thromboplastin time had to be within the therapeutic range of intended use of anticoagulants.
10. Female patients of childbearing potential had to have a negative urine or serum pregnancy test within 72 hours before the first dose of study treatment. If the urine test was positive or could not be confirmed as negative, a serum pregnancy test was required.
11. Patients (both male and female) of reproductive potential had to be willing to practice highly effective methods of contraception throughout the study and for 120 days after the last dose of study treatment. Abstinence was acceptable if this was the usual lifestyle for the patient. Female patients were considered NOT of childbearing potential if they had a history of surgical sterility or evidence of post-menopausal status defined as any of the following:

    1. ≥45 years of age and not having menses for more than 1 year.
    2. Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle stimulating hormone (FSH) value in the post-menopausal range upon Screening evaluation.
    3. Post-hysterectomy, oophorectomy, or tubal ligation; documented hysterectomy or oophorectomy had to be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation had to be confirmed with medical records of the actual procedure.
12. Had resolution of toxic effect(s) of the most recent prior cancer therapy to Grade 1 or less (except alopecia). If patient received major surgery or radiation therapy of >30 Gy, they had to have recovered from the toxicity and/or complications from the intervention.

Exclusion Criteria:

1. Had disease suitable for local therapy administered with curative intent.
2. Had received more than 1 prior line of chemotherapy for advanced or metastatic adenocarcinoma of the lung. For all cohorts: Note: Patients may have received additional prior radiotherapy or chemotherapy in the adjuvant setting, providing it was completed at least 6 months prior to start of study treatment.
3. Cohort A: Had received prior therapy with an immunomodulatory agent; Cohort B: Had received prior chemotherapy alone or in combination with immunotherapy in the metastatic setting.
4. Had a known additional malignancy that was progressing or required active treatment; Note: Exceptions included basal cell carcinoma of the skin, squamous cell carcinoma of the skin that had undergone potentially curative therapy, or in situ cervical cancer.
5. Had known active central nervous system (CNS) metastases and/or carcinomatous meningitis; Note: Patients with previously treated brain metastases could participate provided they were stable (without evidence of progression by scans [using the identical modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurological symptoms had returned to Baseline), having no evidence of new or enlarging brain metastases, and were not using steroids for at least 7 days prior to study treatment.
6. History of the following cardiac conditions:

   1. Congestive cardiac failure of > Grade II severity according to the New York Heart Association (defined as symptomatic at less than ordinary levels of activity).
   2. Ischemic cardiac event including, myocardial infarction, within 3 months before the first dose.
   3. Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (ie, sustained systolic blood pressure (BP) >160 mm Hg or diastolic BP >90 mm Hg), or need to change medication because of lack of disease control within 6 weeks before the provision of consent.
   4. History or presence of sustained bradycardia (≤55 beats per minute), left bundle branch block, cardiac pacemaker, or ventricular arrhythmia; Note: Patients with a supraventricular arrhythmia requiring medical treatment but with a normal ventricular rate were eligible.
   5. Family history of long QTc syndrome, personal history of long QTc syndrome, or previous drug-induced QTc prolongation of at least Grade 3 (QTc >500 msec).
7. Abnormal left ventricular ejection fraction on echocardiography or multigated acquisition scan (MUGA) (less than the lower limit of normal for a patient of that age at the treating institution or <45%, whichever was lower).
8. Current treatment with any agent known to cause Torsades de Pointes which could not be discontinued at least 5 half-lives or 2 weeks prior to the first dose of study treatment.
9. Screening 12-lead electrocardiogram (ECG) with a measurable QTc interval according to Fridericia's correction >450 msec.
10. Was currently participating and receiving study therapy or had participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment.
11. Had participated in a study involving any immune checkpoint inhibitor other than currently approved immune checkpoint inhibitors for their lung cancer.
12. Received chemotherapy or targeted small-molecule therapy or radiation therapy within 2 weeks before starting study treatment or who had not recovered (ie, ≤ Grade 1 at Baseline) from adverse events (AEs) due to a previously administered agent.
13. Received an anti-cancer mAb within 4 weeks prior to the first dose of study treatment or who had not recovered (ie, ≤ Grade 1 or Baseline) from AEs due to agents administered more than 4 weeks earlier.
14. Major surgery within 28 days before start of study treatment and failure to have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of study treatment.
15. Received transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (CSFs) (including granulocyte-CSF, granulocyte macrophage-CSF, or recombinant erythropoietin) within 4 weeks prior to the first dose of study treatment.
16. Had a diagnosis of immunodeficiency or was receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment; Note: The use of physiologic doses of corticosteroids could have been approved after consultation with the Sponsor.
17. Active autoimmune disease that had required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs);
18. Known history of human immunodeficiency virus (HIV 1/2 antibodies).
19. Had known active infection with hepatitis B (eg, hepatitis B surface antigen reactive) or hepatitis C (eg, hepatitis C virus RNA [qualitative] was detected).
20. Had received a live-virus vaccination within 30 days of planned treatment start.
21. Had a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
22. Had a history of interstitial lung disease.
23. Inability to swallow or tolerate oral medication.
24. Existing gastrointestinal disease affecting drug absorption, such as celiac disease or Crohn's disease, or previous bowel resection, which was considered to be clinically significant or could interfere with absorption.
25. Known lactose intolerance.
26. Required vitamin K antagonists.
27. Treatment with any of the following: proton pump inhibitors or antacids within 7 days of the start of the study.
28. Treatment with any medication that was predominantly metabolized by CYP3A4 and had a narrow therapeutic index.
29. Known severe hypersensitivity (≥ Grade 3) to bemcentinib, pembrolizumab, and/or any of their excipients.
30. Any evidence of severe or uncontrolled systemic conditions (eg, severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions or ongoing.
31. Had active infection requiring systemic therapy (apart from cutaneous infections)
32. Had received radiation to the lung of >30 Gy within 6 months of the first dose.
33. Had a history or current evidence of any condition, therapy, or laboratory abnormality that could confound the results of the study, interfere with the patient's participation for the full duration of the study, or mean it was not in the best interest of the patient to participate, in the opinion of the Investigator.
34. Was pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting from Screening through to 120 days after the last dose of study treatment.
35. Had known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
36. Cohorts B and C: Had an EGFR mutation or ALK genomic rearrangement.
37. Had received an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Medical College of Wisconsin, 9200 W Wisconsin Avenue, Milwaukee, Wisconsin
- Radiumhospitalet, Oslo University Hospital PB, Oslo, Norway
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol-ICO, Barcelona, Badalona
  - Hospital Teresa Herrera, A Coruña
  - Servicio de Oncologia Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron (VHIR), Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimene Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Servicio de oncologia, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Christie NHS Hospital Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification [text, tables, figures and appendices].
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposal should be directed to clinical@bergenbio.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Li H, Liu Z, Liu L, Zhang H, Han C, Girard L, Park H, Zhang A, Dong C, Ye J, Rayford A, Peyton M, Li X, Avila K, Cao X, Hu S, Alam MM, Akbay EA, Solis LM, Behrens C, Hernandez-Ruiz S, Lu W, Wistuba I, Heymach JV, Chisamore M, Micklem D, Gabra H, Gausdal G, Lorens JB, Li B, Fu YX, Minna JD, Brekken RA. AXL targeting restores PD-1 blockade sensitivity of STK11/LKB1 mutant NSCLC through expansion of TCF1+ CD8 T cells. Cell Rep Med. 2022 Mar 15;3(3):100554. doi: 10.1016/j.xcrm.2022.100554. eCollection 2022 Mar 15. PMID 35492873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was undertaken with 19 sites across 4 countries. The recruitment process began in October 2017 and concluded in October 2022. A sufficient number of volunteers were screened in order to successfully recruit 99 completing patients.
Pre-assignment Details: Participants were screened to the inclusion/exclusion criteria of the protocol. The following assessments were performed: Informed Consent, Demographics, Medical History, Pregnancy/FSH, ECOG performance score, Vital signs, Physical examination, Laboratory Safety Testing, ECG, Tumour assessment scans/biopsy, disease assessment and biomarker assessment.
Groups:
- Cohort A: Cohort A a safety run- in, enrolled participants who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy of any kind to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Cohort B: Cohort B enrolled participants who received a maximum of one prior line of an anti-PD-(L)1 therapy (monotherapy) to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Cohort C: Cohort C enrolled participants who received a maximum of one prior line of therapy with an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 50 | 29 | 20
Completed | 14 | 7 | 1
Not Completed | 36 | 22 | 19

BASELINE CHARACTERISTICS:
Population: This analysis population included all 99 enrolled participants.
Groups:
- Cohort A: Cohort A enrols participants who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy of any kind to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Cohort B: Cohort B enrols participants who received a maximum of one prior line of an anti-PD-(L)1 therapy (monotherapy) to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Cohort C: Cohort C enrols participants who received a maximum of one prior line of therapy with an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 50 | 29 | 20 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.27) | 64.6 (9.41) | 64.8 (9.33) | 64.4 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 6 | 34
  Male | 30 | 21 | 14 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 27 | 20 | 94
  Asian | 2 | 0 | 0 | 2
  Black | 0 | 2 | 0 | 2
  Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 71.92 (13.296) | 72.61 (17.146) | 76.00 (16.096) | 72.95 (15.003)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) includes all participants who have a partial (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by CT scan or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions,. ORR was defined as the percentage of evaluable patients who had at least 1 confirmed overall response CR or PR according to modified RECIST 1.1 evaluation and definitions of disease response.
Time Frame: The disease response is the best improvement or change in a participants cancer burden, as measured from baseline (screening) and then measured again at regular intervals over the whole period of the study, an average of 24 months.
Population: This analysis population included all 90 participants who received at least 1 combination dose of bemcentinib and pembrolizumab, had measurable disease at study entry, met the inclusion/exclusion criteria, and had at least 1 on-treatment scan.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Cohort A enrolled participants who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy of any kind to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Bemcentinib capsules are administered at 400mg for days 1-3, and 200mg thereafter. Pembrolizumab is an IV infusion, administered at a dose of 200mg every 3 weeks.
- Total Patients: This analysis population included all 90 participants who received at least 1 combination dose of bemcentinib and pembrolizumab, had measurable disease at study entry, met the inclusion/exclusion criteria, and had at least 1 on-treatment scan.
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 44 | 27 | 19 | 90
Participants | 10 | 0 | 0 | 10

2. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate includes all participants who have a partial or complete response, or who maintain stable disease.
Time Frame: Disease response is assessed every 9 weeks for the first 45 weeks and then every 12 weeks until disease progression (worsens) or study completion, an average of 24 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 44 | 27 | 19 | 90
Participants | 24 | 12 | 10 | 46

3. Secondary Outcome: Duration of Response
Description: Duration of response includes participants with a partial or complete response and is measured from the date of response until the cancer progresses (worsens).
Time Frame: Disease response is assessed every 9 weeks for the first 45 weeks and then every 12 weeks until disease progression or study completion, an average of 24 months.
Population: This analysis population included all 10 participants with partial (PR) or complete (CR ) response per Response Evaluation Criteria in Solid Tumours Criteria (RECIST v1.0) for target lesions and assessed by CT scan or MRI.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 10 | 0 | 0 | 10
months | 8.1 [3.9 to 25.6] |  |  | 8.1 [3.9 to 25.6]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from the date of the 1st dose of the 1st cycle until the date of progression (the date on which the progression is initially observed) or the date of death (whichever is earlier).
Time Frame: Disease assessments are conducted at screening and then every 9 weeks for the first 45 weeks and then every 12 weeks until disease progression or death, whichever comes first, up to study completion (an average of 24 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 44 | 27 | 19 | 90
weeks | 35.7 [18.0 to 54.1] | 26.1 [9.6 to 36.0] | 26.0 [9.7 to 64.4] | 27.1 [19.0 to 38.0]

5. Secondary Outcome: Overall Survival
Description: Time to death is measured from the date of first dose until the date of death or the date the participants is last known to be alive. It includes all participants.
Time Frame: Survival visits are conducted every 12 weeks after disease progression until death or until study completion (an average of 24 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 44 | 27 | 19 | 90
weeks | 61.0 [46.3 to 75.9] | 43.7 [29.1 to 70.1] | 64.4 [27.9 to 110.7] | 56.6 [43.7 to 66.7]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants with each adverse event (AE) will be summarized.
Time Frame: Adverse events are collected from the date of consent until up to 120 days after cessation of both treatments, up to 24 months of treatment, followed by an additional 120 days following cessation, up to 27 months total.
Population: This analysis population included all 99 enrolled participants who received at least one dose of study treatment (bemcentinib and pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 50 | 29 | 20 | 99
Participants | 49 | 29 | 20 | 98

7. Secondary Outcome: Pharmacokinetic (PK) Parameters: Maximum Observed Concentration (Cmax)
Description: Cmax defined as the maximum observed concentration. These Cmax results are after the maintenance dose.
Time Frame: Up to 106 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 50 | 29 | 20 | 99
ng/mL | 270 (165) | 304 (153) | 244 (134) | 275 (156)

8. Secondary Outcome: PK Parameters: Area Under the Curve (AUC)
Description: AUC defined as the area under the concentration versus time curve. Measured as AUC 0-24h, area under the concentration versus time curve from time 0 to 24 hours post-dose at steady state following the maintenance dose per cohort.
Time Frame: Cycle 1 Day 1 and Day 3 pre-dose, and 2, 4, 6, 8 hours post-dose; Cycle 1 Day 2 , Day 4 ,Day 8 and Day 15 pre-dose; Cycle 2 Day 1, and Cycle 3 Day 1., pre-dose. Each cycle is 21 days in duration.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 50 | 29 | 20 | 99
ng.h/mL | 6250 (3880) | 7090 (3620) | 5640 (3200) | 6370 (3680)

9. Secondary Outcome: PK Parameters: Elimination Half-life (T½)
Description: T½ defined as the elimination half-life. Measured at steady state following the maintenance dose per cohort.
Time Frame: Up to 106 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort A | Cohort B | Cohort C | Total Patients
Number analyzed (Participants) | 50 | 29 | 20 | 99
hours | 181 (263) | 192 (195) | 135 (89.9) | 175 (218)

10. Secondary Outcome: Frequency of Clinical Laboratory, Vital Signs, and Electrocardiogram (ECG) Abnormalities.
Description: Number of events (Frequency) of clinically significant laboratory (hematology, including coagulation, urinalysis), vital signs (temperature, systolic blood pressure, diastolic blood pressure, heart rate, and respiratory rate), and ECG abnormalities.
Time Frame: Up to 106 weeks
Population: as for outcome 6
Measure: Number; unit: events
Groups:
- Bemcentinib + Pembrolizumab: Cohort A enrols participants who received a maximum of 1 prior line of platinum-containing chemotherapy and no prior immunotherapy of any kind to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Cohort B enrols participants who received a maximum of one prior line of an anti-PD-(L)1 therapy (monotherapy) to receive bemcentinib (BGB324) in combination with pembrolizumab.
  Cohort C enrols participants who received a maximum of one prior line of therapy with an anti-PD-(L)1 therapy in combination with a platinum-containing chemotherapy.
Arm/Group | Bemcentinib + Pembrolizumab
Number analyzed (Participants) | 99
events
  Hematological | 19
  Clinical Chemistry | 289
  Urinalysis | 0
  Vital signs | 0
  ECG | 43

ADVERSE EVENTS:
Time Frame: Up to 106 weeks
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 41/50 | 22/29 | 14/20
Serious Adverse Events (participants affected / at risk) | 29/50 | 11/29 | 9/20
Other Adverse Events (participants affected / at risk) | 21/50 | 18/29 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=50) | Cohort B (N=29) | Cohort C (N=20)
Pneumonia (Infections and infestations) | 5 (6) | 2 (2) | 2 (4)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fecalith (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertransaminasemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (12) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (8) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=50) | Cohort B (N=29) | Cohort C (N=20)
Asthenia (General disorders) | 11 | 7 | 2
Fatigue (General disorders) | 7 | 8 | 7
Pyrexia (General disorders) | 5 | 7 | 4
Influenza like illness (General disorders) | 6 | 2 | 0 (0)
Oedema peripheral (General disorders) | 3 | 4 | 1
Non-cardiac chest pain (General disorders) | 5 | 0 (0) | 1
Peripheral swelling (General disorders) | 0 (0) | 1 | 2
General physical health deterioration (General disorders) | 0 (0) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0 (0)
Pain (General disorders) | 1 | 0 (0) | 1
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1
Chest pain (General disorders) | 1 | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 | 0 (0)
Device related thrombosis (General disorders) | 1 | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1
Hunger (General disorders) | 0 (0) | 0 (0) | 1
Illness (General disorders) | 0 (0) | 0 (0) | 1
Malaise (General disorders) | 0 (0) | 1 | 0 (0)
Suprapubic pain (General disorders) | 1 | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 1
Blood creatinine increased (Investigations) | 11 | 11 | 8
Alanine aminotransferase increased (Investigations) | 10 | 7 | 4
Aspartate aminotransferase increased (Investigations) | 11 | 6 | 6
Electrocardiogram QT prolonged (Investigations) | 6 | 7 | 4
Amylase increased (Investigations) | 3 | 0 (0) | 3
Blood alkaline phosphatase increased (Investigations) | 6 | 2 | 0 (0)
Weight decreased (Investigations) | 3 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 0 (0)
Blood cholesterol increased (Investigations) | 2 | 3 | 0 (0)
Blood bilirubin increased (Investigations) | 1 | 1 | 1
Platelet count decreased (Investigations) | 2 | 2 | 0 (0)
Neutrophil count decreased (Investigations) | 2 | 1 | 0 (0)
Lymphocyte count decreased (Investigations) | 2 | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1
Blood folate decreased (Investigations) | 0 (0) | 1 | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 | 0 (0)
Computerised tomogram abnormal (Investigations) | 0 (0) | 0 (0) | 1
Cortisol decreased (Investigations) | 0 (0) | 1 | 0 (0)
Ejection fraction decreased (Investigations) | 1 | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 | 0 (0) | 0 (0)
Urine bilirubin increased (Investigations) | 1 | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 20 | 12 | 8
Nausea (Gastrointestinal disorders) | 12 | 7 | 5
Vomiting (Gastrointestinal disorders) | 7 | 6 | 4
Constipation (Gastrointestinal disorders) | 7 | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 | 0 (0) | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 (0)
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
Poor dental condition (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
Toothache (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 (0) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 (0) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 | 5 | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 | 0 (0) | 2
Urinary tract infection (Infections and infestations) | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 (0)
Oral candidiasis (Infections and infestations) | 2 | 0 (0) | 1
Candida infection (Infections and infestations) | 1 | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 | 0 (0)
Fungal infection (Infections and infestations) | 1 | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1
Gastroenteritis (Infections and infestations) | 1 | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 | 0 (0) | 0 (0)
Oral herpes zoster (Infections and infestations) | 1 | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 | 0 (0)
Skin candida (Infections and infestations) | 1 | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1
Toxic shock syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1
Decreased appetite (Metabolism and nutrition disorders) | 16 | 9 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 (0) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0 (0) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 (0) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 10 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 2 | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 (0)
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 (0)
Amnesia (Nervous system disorders) | 1 | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1
Memory impairment (Nervous system disorders) | 1 | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1
Insomnia (Psychiatric disorders) | 5 | 1 | 0 (0)
Anxiety (Psychiatric disorders) | 2 | 1 | 0 (0)
Depression (Psychiatric disorders) | 2 | 0 (0) | 1
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 | 0 (0)
Confusional state (Psychiatric disorders) | 1 | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 | 0 (0)
Depressed mood (Psychiatric disorders) | 1 | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 (0) | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 | 0 (0)
Hypertension (Vascular disorders) | 2 | 0 (0) | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 | 0 (0)
Varicose vein (Vascular disorders) | 1 | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 | 0 (0) | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 | 0 (0)
Photopsia (Eye disorders) | 1 | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT03184571/Prot_SAP_001.pdf